CLINICAL TRIAL: NCT07257926
Title: Prevention of Delayed Post-polypectomy Bleeding by Endoscopic Sucralfate Spray in High-risk Patients: A Randomized Controlled Trial
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Principal Investigator, Hsueh-Chien Chiang, Attending Physician, National Cheng-Kung University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: A-BR-114-027
Record Dates: First submitted 2025-10-09; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-10

CONDITIONS: Bleeding After GI Endoscopy
Keywords: polypectomy; sucralfate; antiplatelet; anticoagulant; postpolypectomy bleeding
MeSH Terms: interventions — Sucralfate; Surgical Instruments

STUDY DESIGN:
Intervention Model Description: After allocation, prophylactic clips will be placed on the polypectomy wounds of patients in the Clipping group. In contrast, 3 g of sucralfate powder will be sprayed on the polypectomy wounds of patients in the Sucralfate group. The powder spray aimed for the full coverage of the polypectomy wound. Six sucralfate tablets (500 mg per Weizip tablet; Yung Shin Pharmaceutical Industries, Taichung, Taiwan) were ground to collect 3 g of sucralfate powder. This powder was then delivered through a functional powder delivery system (7F polyethylene catheter in connection by an oxygen cannula to the air source; propelling power: 1 L/min airflow from the hospital's air source, oxygen or CO2)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Clipping group (Active Comparator): After identifying a resectable colon polyp (size ≥ 1 cm), the operator performed a hot polypectomy. Following hot polypectomy, the wound was observed for 30 seconds to detect potential immediate bleeding. Standard endoscopic interventions such as diluted epinephrine injection, heat coagulation, or clipping were promptly administered if immediate bleeding occurred. Subsequently, the patients were randomly assigned to either the Sucralfate or Clipping groups. After allocation, prophylactic clips will be placed on the polypectomy wounds of patients in the Clipping group.
  Interventions: Device: Clip
- Sucralfate group (Experimental): After identifying a resectable colon polyp (size ≥ 1 cm), the operator performed a hot polypectomy. Following hot polypectomy, the wound was observed for 30 seconds to detect potential immediate bleeding. Standard endoscopic interventions such as diluted epinephrine injection, heat coagulation, or clipping were promptly administered if immediate bleeding occurred. Subsequently, the patients were randomly assigned to either the Sucralfate or Clipping groups. After allocation, 3 g of sucralfate powder will be sprayed on the polypectomy wounds of patients in the Sucralfate group. The powder spray aimed for the full coverage of the polypectomy wound. Six sucralfate tablets (500 mg per Weizip tablet; Yung Shin Pharmaceutical Industries, Taichung, Taiwan) were ground to collect 3 g of sucralfate powder. This powder was then delivered through a functional powder delivery system (7F polyethylene catheter in connection by an oxygen cannula to the air source; propelling power: 1 L/min airflow)
  Interventions: Drug: Sucralfate

INTERVENTIONS:
Drug: Sucralfate — 3 g of sucralfate powder will be sprayed on the polypectomy wounds of patients in the Sucralfate group.
  Arms: Sucralfate group
Device: Clip — Prophylactic clips will be placed on the polypectomy wounds of patients in the Clipping group
  Arms: Clipping group

SUMMARY:
Background： Colonoscopy can detect colon polyps and perform excision to the polyps to prevent colon cancer. However, delayed polypectomy bleeding is one of the complications to be noticed, which has an occurrence rate of about 1-2%, especially large polyps over 1cm with hot snare polypectomy. Colonoscopic clipping was applied for the treatment of bleeding. However, prophylactic clipping after polypectomy was not proved to reduce the rate of delayed polypectomy bleeding. Sucralfate is used for peptic ulcer treatment, which can become a protective layer on the wound to prevent environmental injury. Our preliminary data revealed the endoscopic sucralfate spray could reduce the delayed bleeding rate among general populations. Whether sucralfate can prevent polypectomy wounds from delayed bleeding in high-risk polyps is unknown.

Aim： This study aimed to compare the efficacy in reducing delayed bleeding rate between sucralfate administration and prophylactic clipping on high-risk polypectomy wounds.

Method： This is a randomized clinical trial. The study will recruit 160 patients. After randomization, 80 patients will be classified into the Sucralfate group and 80 into the Clipping group. The participants will receive an endoscopic survey as routine, and we will enroll all patients who take antiplatelets or anticoagulants with polyp size ≥ 1 cm after hot snare polyp excision. Exclusion criteria include patients with an allergy to sucralfate. If immediate polypectomy bleeding occurs, we will apply standard endoscopic therapy by either local injection of diluted epinephrine, heater probe coagulation, and/or hemoclipping. After then, we will spray 3g of sucralfate powder through colonoscopy precisely on the polypectomy wound in the Sucralfate group, and prophylactic clipping will be placed on the polypectomy wound in the Clipping group. All enrolled patients will be monitored for delayed bleeding for 28 days after the colonoscopy.

Expected results and clinical importance:

This study is expected to find that the use of sucralfate powder can more effectively reduce the bleeding risk in high-risk wounds compared to prophylactic clips. In addition to promoting the implementation of national health policies and reducing public exposure to the risk of complications, it can also help avoid medical expenses resulting from complications.

DETAILED DESCRIPTION:
Colonoscopic polypectomy is a key procedure for prevention of colorectal cancer and reduction of associated mortality risk. However, this procedure carries a risk of postpolypectomy bleeding. Postoperative bleeding can occur immediately (intraoperatively, manageable during colonoscopy) or after a while (for example, a month after colonoscopy). The causes of delayed postpolypectomy bleeding include detachment of eschar due to stool passage and extension of submucosal necrosis due to hot snare polypectomy. The incidence rate of delayed postpolypectomy bleeding ranges from 1% to 2%; this rate increases to 6% in patients with large (> 2 cm) colon polyps. Risk factors for this complication include hot snare polypectomy, chronic kidney disease, liver cirrhosis, antiplatelet agent or anticoagulant use, and pedunculated colon polyps. Delayed postpolypectomy bleeding is a major complication that requires prompt management. Patients with delayed bleeding usually present with hematochezia, anemia, hemodynamic instability, or end-organ damage. Hemostasis often requires repeated colonoscopic procedures and hospitalization, which increases patient discomfort and treatment costs. In complex cases, emergent surgical intervention or transarterial embolization may become necessary. Therefore, the prevention of delayed postpolypectomy bleeding is crucial for both patients and clinicians.

Sucralfate, a basic aluminum salt of sucrose octa sulfate, has been used in the treatment of gastrointestinal ulcers; this powder accelerates healing and prevents bleeding. The mechanisms underlying its effects involve binding to exposed proteins on damaged cells and creating a protective layer that shields the mucosa from further injury. Sucralfate can also bind to growth factors and thus promote angiogenesis and mucosal healing. Pharmacodynamic insights have suggested that local application of sucralfate is more effective in promoting wound healing than systemic administration, likely because of its ability to locally adhere to damaged mucosa, forming a sticky coating that accelerates healing.

Liquid sucralfate has demonstrated healing efficacy in endoscopic mucosal resection-induced gastric ulcers. Rectosigmoid ulcer lesions can also be treated with topical sucralfate by enema. In radiation proctitis and idiopathic ulcerative proctitis, sucralfate enemas produced clinical and endoscopic improvement. Compared to the drug powder, we think the liquid formulation would soon drain away from the wound. Therefore, we assume that the local application of sucralfate powder to polypectomy wounds would effectively prevent delayed postpolypectomy bleeding.

In our preliminary data of a pilot study (IRB: A-BR-111-085, ClinicalTrials.gov ID: NCT05817656), a total of 160 patients with polyps (size≥0.5cm) who had undergone colonoscopic polypectomy were enrolled. divided into the sucralfate and control groups (80 per group). After polypectomy, the patients received standard treatment for immediate bleeding. Then, they were randomly allocated to either a sucralfate group (prophylactic spraying of 3g sucralfate powder on polypectomy wounds) or a control group. As a result, the rate of delayed postpolypectomy bleeding (0% vs 6.3%, respectively; P=0.029) and postpolypectomy overt bloody stool (2.4% vs 18.8%, respectively; P=0.001) were lower in the sucralfate group than in the control group. The duration of freedom from delayed bleeding was longer in the sucralfate group than in the control group (P=0.024). Colonoscopic spraying of sucralfate powder is a safe approach with potential to reduce the risk of delayed postpolypectomy bleeding among the general population.

However, whether this method can be applied to high-risk polyps were indetermined, such as large polyps > 1cm under hot snare polypectomy, especially in those who take antiplatelets or anticoagulants. Moreover, the prophylactic potency comparison between sucralfate spray and prophylactic clips was also unknown. Therefore, a head-to-head comparison between sucralfate powder and clipping is needed to identify the preventative potency.

ELIGIBILITY:
Inclusion Criteria:

* patients who take antiplatelets or anticoagulants with large polyps (size ≥ 1 cm)

Exclusion Criteria:

* lacked complete data (serum creatinine, platelet count, and prothrombin time) pertaining to the previous 6 months
* those who did not discontinue or inadequately discontinued antiplatelet agents or anticoagulants
* those who had a known allergy to sucralfate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Rate of delayed postpolypectomy bleeding | 28 days
  Delayed postpolypectomy bleeding was defined as the need for reintervention or hospitalization, indicating a clinically significant bleeding event

SECONDARY OUTCOMES:
Rate of overt bloody stool | 2 days
  Overt bloody stool with spontaneous bleeding cessation was regarded as minor bleeding
Rate of severe bleeding from polypectomy wounds | 28 days
  bleeding from polypectomy wounds necessitating transarterial embolization or emergency surgery

IPD SHARING:
Plan to Share IPD: Yes
after publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: after study publication

REFERENCES:
- [Result] Chiang HC, Chen PJ, Yang EH, Kuo TL, Hsieh MT, Kang JW, Cheng HC, Chang WL, Chen WY, Chiu HC, Lin MY, Hong TC, Chiang CM, Chen WC, Huang KK, Lu MH, Wu MH, Chen CY, Lin XZ, Chuang CH. Clinical Trial: Precise Administration of Sucralfate Powder in Prevention of Delayed Postpolypectomy Bleeding. A Randomized Controlled Trial. Clin Transl Gastroenterol. 2025 Apr 1;16(4):e00818. doi: 10.14309/ctg.0000000000000818. PMID 39836033
- [Result] Chiang HC, Chen PJ, Yang EH, Hsieh MT, Shih IC, Cheng HC, Chang WL, Chen WY, Chiu HC, Kuo HY, Tsai WC, Lo YN, Yang KC, Chiang CM, Chen WC, Huang KK, Tseng HH, Chen CY, Lin XZ, Chuang CH. Precise application of topical tranexamic acid to enhance endoscopic hemostasis for peptic ulcer bleeding: a randomized controlled study (with video). Gastrointest Endosc. 2023 Nov;98(5):755-764. doi: 10.1016/j.gie.2023.06.013. Epub 2023 Jun 24. PMID 37356632
- [Result] Ye Z, Reintam Blaser A, Lytvyn L, Wang Y, Guyatt GH, Mikita JS, Roberts J, Agoritsas T, Bertschy S, Boroli F, Camsooksai J, Du B, Heen AF, Lu J, Mella JM, Vandvik PO, Wise R, Zheng Y, Liu L, Siemieniuk RAC. Gastrointestinal bleeding prophylaxis for critically ill patients: a clinical practice guideline. BMJ. 2020 Jan 6;368:l6722. doi: 10.1136/bmj.l6722. PMID 31907223
- [Result] Wang Y, Ye Z, Ge L, Siemieniuk RAC, Wang X, Wang Y, Hou L, Ma Z, Agoritsas T, Vandvik PO, Perner A, Moller MH, Guyatt GH, Liu L. Efficacy and safety of gastrointestinal bleeding prophylaxis in critically ill patients: systematic review and network meta-analysis. BMJ. 2020 Jan 6;368:l6744. doi: 10.1136/bmj.l6744. PMID 31907166
- [Result] Gutta A, Gromski MA. Endoscopic Management of Post-Polypectomy Bleeding. Clin Endosc. 2020 May;53(3):302-310. doi: 10.5946/ce.2019.062. Epub 2019 Sep 17. PMID 31525836
- [Result] Buddingh KT, Herngreen T, Haringsma J, van der Zwet WC, Vleggaar FP, Breumelhof R, Ter Borg F. Location in the right hemi-colon is an independent risk factor for delayed post-polypectomy hemorrhage: a multi-center case-control study. Am J Gastroenterol. 2011 Jun;106(6):1119-24. doi: 10.1038/ajg.2010.507. Epub 2011 Jan 25. PMID 21266961
- [Result] Elliott TR, Tsiamoulos ZP, Thomas-Gibson S, Suzuki N, Bourikas LA, Hart A, Bassett P, Saunders BP. Factors associated with delayed bleeding after resection of large nonpedunculated colorectal polyps. Endoscopy. 2018 Aug;50(8):790-799. doi: 10.1055/a-0577-3206. Epub 2018 Apr 6. PMID 29625506
- [Result] Bendall O, James J, Pawlak KM, Ishaq S, Tau JA, Suzuki N, Bollipo S, Siau K. Delayed Bleeding After Endoscopic Resection of Colorectal Polyps: Identifying High-Risk Patients. Clin Exp Gastroenterol. 2021 Dec 24;14:477-492. doi: 10.2147/CEG.S282699. eCollection 2021. PMID 34992406
- [Result] Rabeneck L, Paszat LF, Hilsden RJ, Saskin R, Leddin D, Grunfeld E, Wai E, Goldwasser M, Sutradhar R, Stukel TA. Bleeding and perforation after outpatient colonoscopy and their risk factors in usual clinical practice. Gastroenterology. 2008 Dec;135(6):1899-1906, 1906.e1. doi: 10.1053/j.gastro.2008.08.058. Epub 2008 Sep 13. PMID 18938166
- [Result] Kim HS, Kim TI, Kim WH, Kim YH, Kim HJ, Yang SK, Myung SJ, Byeon JS, Lee MS, Chung IK, Jung SA, Jeen YT, Choi JH, Choi KY, Choi H, Han DS, Song JS. Risk factors for immediate postpolypectomy bleeding of the colon: a multicenter study. Am J Gastroenterol. 2006 Jun;101(6):1333-41. doi: 10.1111/j.1572-0241.2006.00638.x. PMID 16771958
- [Result] Ferlitsch M, Moss A, Hassan C, Bhandari P, Dumonceau JM, Paspatis G, Jover R, Langner C, Bronzwaer M, Nalankilli K, Fockens P, Hazzan R, Gralnek IM, Gschwantler M, Waldmann E, Jeschek P, Penz D, Heresbach D, Moons L, Lemmers A, Paraskeva K, Pohl J, Ponchon T, Regula J, Repici A, Rutter MD, Burgess NG, Bourke MJ. Colorectal polypectomy and endoscopic mucosal resection (EMR): European Society of Gastrointestinal Endoscopy (ESGE) Clinical Guideline. Endoscopy. 2017 Mar;49(3):270-297. doi: 10.1055/s-0043-102569. Epub 2017 Feb 17. PMID 28212588
- [Result] Hsu WF, Chang CY, Chang CC, Chang LC, Chen CH, Lin CC, Lin YM, Lee CL, Wu HY, Lee HC, Lee YC, Su MY, Lin LJ, Chia SL, Wu MS, Chiu HM; Colonoscopy Quality Assurance Joint Working Group of Taiwan Colorectal Cancer Screening Program and Digestive Endoscopy Society of Taiwan. Risk of colonoscopy-related complications in a fecal immunochemical test-based population colorectal cancer screening program. Endoscopy. 2022 Mar;54(3):290-298. doi: 10.1055/a-1328-5126. Epub 2021 Feb 24. PMID 33271603
- [Result] Zauber AG, Winawer SJ, O'Brien MJ, Lansdorp-Vogelaar I, van Ballegooijen M, Hankey BF, Shi W, Bond JH, Schapiro M, Panish JF, Stewart ET, Waye JD. Colonoscopic polypectomy and long-term prevention of colorectal-cancer deaths. N Engl J Med. 2012 Feb 23;366(8):687-96. doi: 10.1056/NEJMoa1100370. PMID 22356322